CLINICAL TRIAL: NCT00353964
Title: A Multi-Center, Randomized, Double Masked, Placebo and Active Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of rEV131 2.5 Mg/mL, rEV131 1.25 Mg/mL, rEV131 0.625 Mg/mL, for the Treatment of Ocular Inflammation After Cataract Surgery
Brief Title: Safety and Efficacy Study of rEV131 in the Treatment of Ocular Inflammation After Cataract Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evolutec Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: EVOL-PRO-06-024
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2006-07

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — rEV131 protein, tick

INTERVENTIONS:
Drug: rEV131
Drug: Prenisolone sodium phosphate 1.0%
Drug: rEV131 vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of three concentrations of rEV131, a new investigational anti-inflammatory agent, compared to placebo (an inactive substance) and an FDA approved anti-inflammatory agent in patients with ocular inflammation who have undergone cataract extraction with intra-ocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* be male or female who has undergone unilateral cataract extraction by phacoemulsification (PHACO) method with implantation of a posterior chamber intraocular lens

Exclusion Criteria:

* have unstable glaucoma
* have an active bacterial and/or viral infection
* use any ocular or systemic anti-inflammatory agents within 1 week prior to enrollment and for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Wynne Weston-Davies, MD, Study Director — Evolutec Group
Locations (1):
- ORA Study Sites, North Andover, Massachusetts, United States